CLINICAL TRIAL: NCT02054000
Title: Effectiveness of Intracoronary Tirofiban on No-Reflow Phenomena in Patients With ST-Elevated Myocardial Infarction Undergoing Primary Percutaneous Coronary Intervention
Brief Title: Intracoronary Tirofiban on No-Reflow Phenomena
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: TC Erciyes University (Other)
Responsible Party: Principal Investigator, Mahmut Akpek, Medical doctor of Cardiology department, TC Erciyes University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Makpek-2
Record Dates: First submitted 2014-01-30; First posted 2014-02-04 (Estimated); Last update posted 2014-02-04 (Estimated); Status verified 2014-02

CONDITIONS: No-Reflow Phenomenon
Keywords: No-reflow phenomenon, tirofiban, intracoronary
MeSH Terms: conditions — No-Reflow Phenomenon | interventions — Tirofiban

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor

ARMS (2):
- Tirofiban group (Active Comparator): If thrombolysis in myocardial infarction flow <3 in spite of performed treatments, patients were considered as no-reflow and randomized to tirofiban or placebo group. Intracoronary tirofiban (25 µgr/kg) was administered via the guiding catheter to the infarct related artery
  Interventions: Drug: Tirofiban
- Placebo group (Placebo Comparator): If thrombolysis in myocardial infarction flow <3 in spite of performed treatments, patients were considered as no-reflow and randomized to tirofiban or placebo group. Intracoronary serum physiologic as placebo was administered via the guiding catheter to the infarct related artery
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Tirofiban — Intracoronary administering of Tirofiban
  Other Names: Glycoprotein IIb/IIIa inhibitor
  Arms: Tirofiban group
Other: Placebo — Intracoronary serum physiologic
  Arms: Placebo group

SUMMARY:
The goal of this study was to evaluate the acute effect of intracoronary administration of tirofiban on no-reflow phenomenon in patients with STEMI and occurrence of no-reflow phenomenon undergoing primary percutaneous coronary intervention (PCI).

DETAILED DESCRIPTION:
The no-reflow phenomenon is one of the most common causes of adverse cardiovascular events in patients with ST-elevated myocardial infarction (STEMI). Re-canalization of infarct related arterial (IRA) flow related to better ventricular performance and lower mortality rate in patients with STEMI. In addition, no-reflow phenomena may limit the benefits of re-canalization of the IRA.

In recent years, many mechanical or pharmacological treatment strategies including adjunctive administration of glycoprotein IIb/IIIa inhibitors (GPI) have been proposed in patients with STEMI. Although current guidelines recommend that small molecule GPI should be administered as an upstream bolus followed by a continuous infusion in patients with STEMI, changes in clinical practice may obviate the need for GPI dosage or routes in current practice. Previous studies have shown that intravenous and intracoronary administration of GPI improve the prognosis and significantly reduce mortality in patients with STEMI. Recently, the Ongoing Tirofiban in Myocardial infarction Evaluation-2 (ON-TIME 2) trial found that the use of tirofiban started during the pre-hospital phase as upstream therapy for primary percutaneous coronary intervention (PCI) and continued for up to 18 hours infusion after the procedure showed an improvement in the markers of reperfusion. Additionally, a reduction was demonstrated in the death in recurrent myocardial infarction in urgent target vessel revascularization and thrombotic bailout. However, in the current literature there are insufficient data regarding the role of intracoronary administration of GPI inhibitors in patients with STEMI who developed the no-reflow phenomenon. The goal of this study was to evaluate the acute effect of intracoronary administration of tirofiban on no-reflow phenomenon in patients with STEMI and occurrence of no-reflow phenomenon undergoing primary PCI.

ELIGIBILITY:
Inclusion Criteria:

- Patients with ST-elevated myocardial infarction who developed no-reflow phenomena

Exclusion Criteria:

* Treatment with thrombolytic drugs in the previous 24 hours
* Known malignancy
* Pain to balloon time >6 hours
* Uncontrolled hypertension (>180/110 mmHg)
* Bleeding diathesis
* Thrombocytopenia
* End-stage liver disease
* Cardiogenic shock
* Renal failure
* Life expectancy of less than 1 year
* Contraindication for the use of tirofiban.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 162 (Actual)
Dates: Start 2011-01; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
in-hospital mortality | up to 8 days
Non-fatal myocardial infarction | up to 8 days
in-stent thrombosis | up to 8 days

CONTACTS AND LOCATIONS:
Locations (1):
- Erciyes University School of Medicine, Kayseri, Turkey (Türkiye)